CLINICAL TRIAL: NCT04490928
Title: The Problem of Incomplete Myocardial Revascularization in Percutaneous Coronary Intervention in Patients With Acute Coronary Syndrome Non-ST-elevation
Brief Title: The Problem of Incomplete Myocardial Revascularization in Percutaneous Coronary Intervention in Patients With NSTEMI
Acronym: CONTRAST
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: 10-19/19
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: NSTEMI
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- complete revascularization: All patients who underwent complete myocardial revascularization
- incomplete revascularization: All patients who did not complete myocardial revascularization
- without revascularization: All patients who were not revascularized

SUMMARY:
The study included all patients admitted to the intensive care unit of the district hospital and sent to the angiographic Department for diagnosis and performance of PCI with a diagnosis of NSTEMI, including myocardial infarction (mi) and unstable angina, determined by clinical data, ECG signs and laboratory indicators. Data from patients living in the Sergiev Posad municipal district will be analyzed in order to achieve maximum registration of adverse events during one year of follow-up.

DETAILED DESCRIPTION:
Objective: to investigate the problem of incomplete myocardial revascularization in percutaneous coronary interventions in patients with acute coronary syndrome without St segment elevation who were admitted to the angiographic Department of the Sergiev Posad city hospital in the Moscow region.

The study will include all patients admitted to the intensive care unit of the regional hospital and sent to the angiographic Department for diagnosis and performance of PCI with acute coronary syndrome NSTEMI, including myocardial infarction (mi) and unstable angina, determined by clinical data, ECG signs and laboratory indicators. Anamnestic, clinical, biochemical indicators, cardiovascular risk factors, comorbid index that determines the course of acute coronary syndrome and prognosis (grace), a number of angiographic data, including the number of affected arteries and variants of the index "syntax score 50" and modified "syntax score 30", "syntax score 70" and" syntax score 90" to separate complete and incomplete revascularization, an integral indicator of the quality of the remaining index Syntex, the absolute value of which is corrected during data analysis. The data of patients living in the city of Sergiev Posad will be reviewed in such a way as to minimize the subsequent year of follow-up, using a telephone survey and the EMIAS electronic system

ELIGIBILITY:
Inclusion Criteria:

- All patients who were referred to an angiographic unit with a diagnosis of NSTEMI for diagnostic coronary angiography and/or PCI from November 2018 to February 2019.

Exclusion Criteria:

* Patients with myocardial infarction with ECG- confirmed ST elevation of more than 1 mm in two leads.
* Residents of areas other than the area in question that may be difficult to contact.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were admitted to the intensive care unit of the district hospital from November 2018 to February 2019 and sent to the angiographic Department for diagnosis and performance of PCI with a diagnosis of NSTEMI, including myocardial infarction (mi) and unstable angina, determined by clinical data, ECG signs and laboratory indicators. Data from patients living in the Sergiev Posad municipal district will be analyzed in order to achieve maximum registration of adverse events during one year of follow-up. (Included in the registry profile)
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Time to non- fatal myocardial infarction, stroke, repeated hospitalizations for cardiovascular reasons, repeated PCI, CABG, cardiovascular death or death from all-cause | 12 months
  Primary Outcome Measures will be evaluated 12 months after the patient is discharged from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Mazaev, Study Director — National Research Center for Therapy and Preventive Medicine
Locations (1):
- Sergiyev Posad city hospital, Sergiyev Posad, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: No